CLINICAL TRIAL: NCT06680492
Title: The Role of Nutrition in Muscle Function of Bariatric Surgery Patients
Status: Recruiting | Type: Observational
Sponsor: Concordia University, Montreal (Other)
Collaborators: Montreal General Hospital (Other)
Responsible Party: Principal Investigator, Sylvia Santosa, Professor, Concordia University, Montreal
Other Study IDs: 90000088
Record Dates: First submitted 2024-10-20; First posted 2024-11-08 (Actual); Last update posted 2024-11-08 (Actual); Status verified 2024-10

CONDITIONS: Obesity, Diabetes, Nutrition, Physical Health; Body Composition Changes; Muscle Function, Handgrip Strength Test; Protein Metabolism; Bariatric Surgery Patients
Keywords: Obesity; Bariatric sugery; Protein function; Muscle function; 6-Minute Walk Test; Handgrip Strength Test; Nutritional needs; Nutritional guides; Nutrition
MeSH Terms: conditions — Obesity; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Blood and urine samples for the purpose of further laboratory analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Current recommendations for protein intake after bariatric surgery are not based on strong scientific evidence. It remains unclear how much protein should be eaten to minimize muscle loss and preserve the metabolism and function of individuals post-bariatric surgery.

The objective of this study is to analyze the relationships between changes in body composition, nutrition and protein intake, and muscle function after bariatric surgery to further our understanding of the nutritional needs of patients after bariatric surgery.

We intend to recruit around 75 participants, men and women, aged between 18 and 65 years. Participants will be recruited from the Bariatric Surgery Clinic, McGill University Health Center.

ELIGIBILITY:
Inclusion Criteria:

* Male and female
* Aged 18 to 65 years old
* Undergoing first bariatric surgery (any type)
* Diabetics and non-diabetics
* Non-smokers and non-cannabis consumers

Exclusion Criteria:

* Pregnant and breastfeeding women
* Individuals undergoing second bariatric surgery
* Regular smokers and cannabis consumers
* Current use of Ozempic (or Ozempic-like medication) and anti-psychotic meds
* Limited physical mobility (using walking aids such as canes, walkers, or wheelchairs) and issues with hand resistance
* Kidney disease, non-controlled / unstable hypertension and hypothyroidism, and any metabolic disease other than diabetes

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Individuals living with obesity to undergo primary bariatric surgery from the Montreal area. Individuals to be recruited from the Montreal General Hospital Bariatric Clinic.
Sampling Method: Non-Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2017-06-23 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Change in weight | Baseline (pre-operation), and at 3-months and 6-months post-operation.
  Overall weight loss (kg)
Change in BMI | Baseline (pre-operation), and at 3-months and 6-months post-operation.
  Height and weight will be measured and combined to report BMI (kg/m^2).
Change in fat mass | Baseline (pre-operation), and at 3-months and 6-months post-operation.
  Body composition is measured by dual-energy x-ray absorptiometry.
Change in overall body fat percentage | Baseline (pre-operation), and at 3-months and 6-months post-operation.
  Body composition is measured by dual-energy x-ray absorptiometry.
Resting Energy Expenditure | Baseline (pre-operation), and at 3-months and 6-months post-operation.
  Resting energy expenditure will be measured in a fasted state by indirect calorimetry. The volume of oxygen and carbon dioxide and water vapor pressure will be taken into consideration to calculate the resting energy expenditure.
Substrate Oxidation | Baseline (pre-operation), and at 3-months and 6-months post-operation.
  Substrate oxidation will be measured in a fasted state by indirect calorimetry. The volume of oxygen, carbon dioxide, and water vapor pressure will be taken into consideration to calculate the respiratory exchange ratio.
Nurition and Protein Intake | Baseline (pre-operation), and at 3-months and 6-months post-operation.
  A 3-day food journal and a 24-hour food recall will measure the nutritional profile (protein intake). A 24-hour urine sample will be used to measure urinary nitrogen concentration.
Hormone and Inflammatory Marker Assays | Baseline (pre-operation), and at 3-months and 6-months post-operation.
  The inflammatory cytokines, chemokines, and adipokines in blood will be measured using Enzyme-Linked Immunosorbent Assay (ELISA).

CONTACTS AND LOCATIONS:
Locations (1):
- Montreal General Hospital (MUHC), Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No